CLINICAL TRIAL: NCT04709744
Title: Impact of Vitamin D Level and Supplement on SLE Patients During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Yasmin Adel Abdelsalam Hussein, Lecturer of Rheumatology and Rehabilitation, Mansoura University
Other Study IDs: RP.21.01.91
Record Dates: First submitted 2021-01-09; First posted 2021-01-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample for Vitamin D level by ELISA
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SLE patients: SLE patients were presented to chest outpatient clinic and emergency hospital, Mansoura University with manifestation suggesting COVID-19 infection. Vit D was measured in serum by ELISA. Vit D was added to anti COVID-19.
  Interventions: Drug: Vitamin D; Diagnostic Test: ELISA

INTERVENTIONS:
Drug: Vitamin D — Impact of serum vit D level in SLE patients with COVID-19 disease on severity of infection, duration of COVID-19 disease course, fatigue development as a complication for both SLE and COVID-19 and assess impact of prior chloroquine on COVID-19 disease outcomes
  Other Names: Serum Vitamin D level
Diagnostic Test: ELISA — Measure vitamin D level

SUMMARY:
Aim of the work Impact of serum vit D level in SLE patients with COVID-19 disease on severity of infection, duration of COVID-19 disease course, fatigue development as a complication for both SLE and COVID-19 and assess impact of prior chloroquine on COVID-19 disease outcomes Patients and methods 38 SLE patients previously diagnosed and on different lines of lupus management. Participants were presented to chest outpatient clinic and emergency hospital, Mansoura University with manifestation suggesting COVID-19 infection. Serum vit D was measured in serum by ELISA.

DETAILED DESCRIPTION:
Primary objective: assess the impact of serum vit D level in SLE patients with COVID-19 disease on severity of infection and pandemic treatment outcome.

Secondary objectives:

* Effect of serum vit D level in SLE patients on duration of COVID-19 disease course and fatigue development as a complication for both SLE and COVID-19
* Impact of prior chloroquine on COVID-19 disease outcomes
* Correlation of serum vit D level with different laboratory investigations at time of COVID-19 outbreak

ELIGIBILITY:
Inclusion Criteria:

* - SLE patients previously diagnosed
* Patients are not suffering from malignancies.
* Patients have no organ failure nor uncontrolled medical illness.
* Recent COVID-19 infection

Exclusion Criteria:

* - Pregnant, lactating females
* Concurrent malignancies
* Patients with other autoimmune disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients infected with COVID-19
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Level of serum vitamin D in SLE infected with COVID-19 | 6 months
  Measurement of serum vit D level (ng/ml)

SECONDARY OUTCOMES:
Vitamin D level with COVID-19 severity | 6 months
  Level of serum vitamin D (ng/ml) in mild, moderate and sever COVID-19

OTHER OUTCOMES:
Impact of serum vit D level in SLE patients on duration of COVID-19 disease course | 6 months
  serum vit D level (ng/ml) in SLE patients and time to recovery (number of days) from COVID-19
Impact of prior chloroquine on COVID-19 disease outcomes | 6 months
  Can prior chloroquine in SLE patients affect outcome of COVID-19 infection (recovery or die)
Serum vitamin D level and development of fatigue | 6 months
  Basal vitamin d level (ng/ml) in SLE patients diagnosed with recent COVID-19 and development of fatigue after recovery from COVID-19 infection
Correlation of serum vit D level with different laboratory investigations at time of COVID-19 outbreak | 6 months
  Correlation of serum vit D level (ng/ml) with ESR, CRP, serum Lymphocyte count, Ferritine, D-dimer at time of COVID-19 diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: yasmin ElbaiomyAdel, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No